CLINICAL TRIAL: NCT04574076
Title: A Multinational, Prospective, Open Labelled, Non-controlled, Non-interventional Post-authorisation Study of Turoctocog Alfa Pegol (N8-GP) During Long-term Routine Prophylaxis and Treatment of Bleeding Episodes in Patients With Haemophilia A
Brief Title: A Study Following Males With Haemophilia A on Prophylaxis With Esperoct®
Acronym: pathfinder9
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7088-4029; EUPAS36536 (Registry Identifier: EU PAS Register); U1111-1235-6007 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-09-21; First posted 2020-10-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- N8-GP: Patients with haemophilia A
  Interventions: Drug: Turoctocog alfa pegol (N8-GP)

INTERVENTIONS:
Drug: Turoctocog alfa pegol (N8-GP) — Patients will be treated with commercially available N8-GP for prophylaxis and treatment of bleeding episodes according to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available N8-GP has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.

SUMMARY:
This study will collect information on side effects and how well Esperoct® (turoctocog alfa pegol (N8-GP)) works during long-term treatment (prophylaxis) in males with haemophilia A. Participants in this study will get the same treatment as they would normally get, if they were not participating in the study. All visits at the clinic are done in the same way as participants are used to, when visiting their doctor. During visits at the clinic participants might be asked for some relevant tests if considered useful by the study doctor. During the visits the study doctor might ask if participants had any side effects since the last study visit. Participants will be asked to note down in their own diary the number of bleeds and how these were treated, as well as their regular prophylaxis. Participation in the study will last for about 5-7 years, depending on when participants join the study. Participants are free to leave the study at any time and for any reason. This will not affect their current and future medical care.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available Esperoct® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.
* Male patients of all ages, according to local label, are allowed in this study
* Diagnosis of severe or moderate Haemophilia A

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Known or suspected hypersensitivity to N8-GP or related products
* Mental incapacity, unwillingness or language barriers precluding adequate understanding and cooperation
* Clinical suspicion or presence of FVIII inhibitors at time of inclusion

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haemophilia A
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2027-06-03 (Estimated); Study Completion 2027-06-03 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) reported during the study period | From inclusion of the patient (Visit 1) until the end of study (Visit 3), duration 5-7 years
  Count of events

SECONDARY OUTCOMES:
Number of Serious Adverse Events (SAEs) reported during the study period | From inclusion of the patient (Visit 1) until the end of study (Visit 3), duration 5-7 years
  Count of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (1452), Study Director — Novo Nordisk A/S
Locations (25):
- AKH - Klin. Abt. f. Haematologie u. Haemostaseologie, Vienna, Austria
- UMHAT "Tsaritsa Yoanna-ISUL", Sofia, Bulgaria
- KBC Zagreb, Rebro, Hemofilija centar, Zagreb, Croatia
- Czechia (2):
  - FN Brno odd. hematologie, Brno
  - FN HK - IV. Interni hematologicka klinika, Hradec Králové
- Estonia (2):
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital Haematology Clinic, Tartu
- Germany (2):
  - Vivantes Netzwerk für Gesundheit GmbH - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitätsklinikum Bonn - Institut für Experimentelle Hämatologie, Bonn
- Greece (2):
  - "Laiko" General Hospital of Athens, Athens
  - Aghia Sophia Childrens' Hospital, Athens
- MH Eü. Központ -Orszagos Haemophilia Kozpont, Budapest, Hungary
- Italy (4):
  - Azienda Ospedaliera-Universitaria Parma, Parma
  - Policlinico Umberto I Sezione Ematologia, Roma
  - A.O.U Città Salute Scienza Torino, Torino
  - Ospedale San Bortolo, Vicenza
- Lithuania (3):
  - Hospital of LUHS "Kauno Klinikos", Kaunas
  - Republican Panevezys Hospital, Public consultation clinic, Panevezys
  - Vilnius University hospital Santaros klinikos, Vilnius
- Portugal (2):
  - Centro Hospitalar Lisboa Norte-HSM, Lisbon
  - ULS São João, E.P.E., Porto
- Unilabs Slovensko, s. r. o., Košice, Slovakia
- PeK - University Children's Hospital, Department of haematology, Ljubljana, Slovenia
- Hospital Regional Universitario de Málaga, Málaga, Spain
- Kinderspital Hämatologie, Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com